CLINICAL TRIAL: NCT00209378
Title: Citrate Versus Heparin Anticoagulation in Continuous Venovenous Hemofiltration in Critically Ill Patients With Acute Renal Failure: A Randomized Clinical Trial
Brief Title: Citrate Versus Heparin Anticoagulation in Continuous Venovenous Hemofiltration
Acronym: CASH-CVVH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Free University Medical Center (Other)
Collaborators: Dirinco B.V. (Industry)
Responsible Party: Principal Investigator, S.A. Nurmohamed, internist-nephrologist, Free University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03.187
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Acute Kidney Injury
Keywords: Continuous venovenous hemofiltration (CVVH); Continuous renal replacement therapy (CRRT); Acute Kidney Injury; Regional citrate anticoagulation; filter survival; trisodium citrate; bleeding complication; Hemofiltration
MeSH Terms: conditions — Acute Kidney Injury | interventions — Citric Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- heparin (Active Comparator): Citrate regional anticoagulation is compared with standard systemic heparinization.
  Interventions: Other: regional anticoagulation with citrate
- Citrate (Active Comparator): regional anticoagulation with citrate containing replacement solution
  Interventions: Other: HfCitPre

INTERVENTIONS:
Other: regional anticoagulation with citrate — Regional anticoagulation with trisodium citrate is compared with standard systemic heparinization.
  Other Names: HFCitPre
  Arms: heparin
Other: HfCitPre — regional anticoagulation with citrate containing replacement solution
  Arms: Citrate

SUMMARY:
The purpose of this study is to compare citrate regional anticoagulation with systemic heparinization in continuous venovenous hemofiltration. The investigators' hypothesis is, that regional citrate anticoagulation with replacement solution containing trisodium citrate, will be associated with lower mortality and less bleeding complications compared to heparin, with also a better filter survival.

DETAILED DESCRIPTION:
Acute renal failure occurs in about 20% of critically ill patients and is associated with increased morbidity and mortality, in spite of modern renal replacement techniques. The latter include continuous venovenous hemofiltration (CVVH) techniques, necessitating anticoagulation of blood entering the extracorporeal circuit to prevent premature clot formation and hemofilter dysfunction. Heparin is commonly used for that purpose, but carries a serious risk of bleeding complications and heparin induced thrombocytopenia. In a subgroup of critically ill patients systemic anticoagulation is absolutely contraindicated. Citrate-anticoagulant CVVH carries the potential advantage of less bleeding complications and prolonged filter survival, but carries the risk of hypocalcaemia, when citrate is inappropriately or insufficiently counteracted by calcium infusion after passage of blood through the filter. In addition, when too much citrate enters the circulation, a metabolic alkalosis may develop, since citrate is converted to bicarbonate by the liver.

Moreover, continuous filtration techniques may attenuate a potentially harmful exaggerated immune response, particularly when high volume filtration (> 6 L/h) is used. Also, the type of anticoagulation may modulate immune responses, as known from biocompatibility studies in intermittent hemodialysis.

In the first part of the research proposal concerning high bleeding risk patients a comparison will be made in a prospective sequential cohort study between no anticoagulation and citrate regarding filter survival time, bleeding risk, dialyser efficacy, circulating immune mediators (such as neutrophil elastase and myeloperoxidase, interleukins, platelet-activating factors, activated complement products, soluble cytokine receptors and adhesion molecules), metabolic balance, and acute renal failure duration. Also, filter survival time will be assessed. The purpose of the second part of the current research proposal is to evaluate in a randomised controlled clinical trial in 350 critically ill patients (18-80 years) with acute renal failure, (2 arms of 175 patients), without an increased bleeding risk (thrombocytes > 40 x 10^9/L, APTT < 60 sec, PT-INR < 2) whether citrate CVVH is better than bicarbonate-heparin CVVH in terms of the same parameters as in the first part of the study but with the addition of mortality as the primary endpoint.

For this purpose a simple predilution system and citrate adjustment protocol will be used and compared to standard heparin dosing. This replacement solution shall be custom made, containing trisodium citrate, no lactate or bicarbonate, no calcium and a low sodium content.

Main objective: Investigation of the mortality during continuous venovenous hemofiltration with systemic anticoagulation with heparin compared with regional anticoagulation with trisodium citrate and also the investigation of the filter survival. Our hypothesis is, that regional citrate anticoagulation with replacement solution containing trisodium citrate, will be associated with less bleeding complications compared to heparin, with also a better filter survival. Most important we want to evaluate the hypothesis that treatment with citrate will result in a lower mortality compared to treatment with systemic heparinization.

Regional anticoagulation with trisodium citrate may also have some potential effects on the immune response as known from biocompatibility studies in intermittent hemodialysis. Bioincompatibility leads to polymorphonuclear cell degranulation as indicated by the release of intracellular granule products such as myeloperoxidase, lactoferrin, lysozyme and elastase. Citrate anticoagulation may lead to a lower polymorphonuclear cell degranulation, since cations play a pivotal role in the process of cell activation and citrate creates an almost calcium-free environment within the dialyser by its virtue to chelate calcium.

Primary endpoints:

Mortality at day 28 after inclusion will be evaluated. Survival time of the first hemofilter used will be determined, including the cause of filter termination and the number of filters used in the first 72 hours; the average filter patency time will be calculated.

Citrate CVVH is stopped and thus also the study, if the patient fulfils one of the following criteria:

1. Total to ionised calcium ratio of more than 2.5.
2. Persistent metabolic alkalosis with a B.E. of more than 10.
3. Clinical signs of hypocalcaemia: tetanic symptoms or prolonged QT interval
4. Progressive non-lactic acidosis (pH < 7.20) during CVVH combined with an increase in anion gap (> 13) without the presence of endo- or exogenous acids other than citrate suggesting citrate accumulation

Patients on heparin developing a HIT will continue CVVH with danaparoid anticoagulation. Patients on heparin developing a bleeding episode will continue CVVH with regional citrate anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted on the Intensive Care Unit (ICU) requiring continuous venovenous hemofiltration.
* No high bleeding risk. A high bleeding risk is defined as a platelet count below 40 x 10^9/L or APTT of more than 60 seconds or a PT-INR of more than 2.0 or a recent major bleeding or significant active bleeding i.e. requirement for more than two units of packed red blood cells as a transfusion within 24 hours of initiation of CVVH.

Exclusion Criteria:

* Less than 18 or over 80 years of age.
* Patients administered heparin or coumarins for other reasons will also be excluded.
* Patients with a HIT in known history will also be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2005-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Mortality | Day 28 after ICU admission

SECONDARY OUTCOMES:
Laboratory markers of inflammation, endothelial dysfunction and coagulation | 72 hours
Filter life (first filter and total amount of filters in 72 hours) | 72 hours
Bleeding complications | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Piet M ter Wee, MD, PhD, Study Director — Amsterdam UMC, location VUmc; Johan Groeneveld, MD, PhD, Study Director — Amsterdam UMC, location VUmc; Shaikh A Nurmohamed, MD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (9):
- Netherlands (9):
  - Medical Center Alkmaar, Alkmaar
  - Slotervaart Ziekenhuis, Amsterdam
  - St Lucas Andreas Ziekenhuis, Amsterdam
  - Vrije Universiteit Medical Center, Amsterdam
  - Rijnstate, Arnhem
  - UMC Groningen, Groningen
  - Spaarne Hospital Hoofddorp, Hoofddorp
  - Rijnland Hospital, Leiderdorp
  - Haga Hospital, The Hague

REFERENCES:
- [Background] Nurmohamed SA, Vervloet MG, Girbes AR, Ter Wee PM, Groeneveld AB. Continuous venovenous hemofiltration with or without predilution regional citrate anticoagulation: a prospective study. Blood Purif. 2007;25(4):316-23. doi: 10.1159/000107045. Epub 2007 Aug 14. PMID 17700015
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078
- [Derived] Schilder L, Nurmohamed SA, Bosch FH, Purmer IM, den Boer SS, Kleppe CG, Vervloet MG, Beishuizen A, Girbes AR, Ter Wee PM, Groeneveld AB; CASH study group. Citrate anticoagulation versus systemic heparinisation in continuous venovenous hemofiltration in critically ill patients with acute kidney injury: a multi-center randomized clinical trial. Crit Care. 2014 Aug 16;18(4):472. doi: 10.1186/s13054-014-0472-6. PMID 25128022
- [Derived] Aman J, Nurmohamed SA, Vervloet MG, Groeneveld AB. Metabolic effects of citrate- vs bicarbonate-based substitution fluid in continuous venovenous hemofiltration: a prospective sequential cohort study. J Crit Care. 2010 Mar;25(1):120-7. doi: 10.1016/j.jcrc.2009.02.013. Epub 2009 May 8. PMID 19427760